CLINICAL TRIAL: NCT06486896
Title: Effect of Adding Interferential Current to Pelvic Floor Muscle Training on Vaginismus: A Randomized Controlled Trial
Brief Title: Effect of Adding Interferential Current to Pelvic Floor Muscle Training on Vaginismus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004953
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Vaginismus
Keywords: Interferential, pelvic floor training, vaginismus
MeSH Terms: conditions — Vaginismus | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor training (Active Comparator): The patients will receive pelvic floor training exercise+ advice 3 times/weekly for 8 weeks
  Interventions: Other: Pelvic floor training; Behavioral: General advice
- Interferential current (Experimental): Patients will receive interferential current+pelvic floor training+advice
  Interventions: Other: Pelvic floor training; Device: Interferential current; Behavioral: General advice

INTERVENTIONS:
Other: Pelvic floor training — It will be in the form of pelvic floor relaxation with biofeedback, as well as stretching exercises for the pelvic floor and the adjacent muscles. The patient will be asked to lie in a comfortable crock lying position. She will be instructed to do diaphragmatic breathing exercises. The vaginal electrode of the biofeedback will be gently introduced into the vagina to start pelvic floor relaxation training. Then, the patient will be asked to perform pelvic floor relaxation by slightly contracting the pubococcygeus muscle. After 10 minutes of pelvic floor relaxation training, the patient will then be instructed to return to the active state gradually, the treatment procedure will be performed 3 times/ week for 8 weeks. Stretching exercises for the pelvic floor and the adjacent muscles: Levator ani & perineal muscles stretch, hip adductor muscles stretch, piriform muscle stretch, hip flexor muscles stretch, and obturator internus muscle stretch.
Device: Interferential current — Each female in the experimental group will receive interferential current, 3o minutes per session, 2 sessions per week, for 8 weeks. The applied parameters will be a frequency of 2000Hz, a modulated amplitude of frequency of 80Hz, pulse width of 200μs, and the intensity is modulated according to the sensory level of each participant. While the participant is in a comfortable crock lying position with abducted hips, the position of the electrodes will be maintained in all sessions
  Arms: Interferential current
Behavioral: General advice — The patients in both groups will follow general advice to help vaginismus for 8 weeks

SUMMARY:
This study aims to determine the effect of adding interferential current to pelvic floor muscle training on vaginismus.

DETAILED DESCRIPTION:
Vaginismus is a common sexual problem with a prevalence of 20% in Egyptian women, that has a significant impact on a person's life, affecting their physical, emotional, and psychological well-being, as well as their relationships and overall quality of life.

There were previous studies that studied the effect of pelvic floor rehabilitation on vaginismus and found that there was a highly significant decrease in pain and pelvic floor muscle spasms, as well as a highly significant increase in sexual function. Also, only one previous protocol explored the effect of interferential current on treating vaginismus. But, till now, there is no prior study that investigated the impact of adding interferential current to pelvic floor muscle training on treating vaginismus. this trial has two groups; one will receive interferential current, and the other group will receive interferential current + pelvic floor muscle training

ELIGIBILITY:
Inclusion Criteria:

1. Women suffer from primary vaginismus with a duration of marriage ranging from 1 to 12 months. They are diagnosed and referred by the gynecologist.
2. Their pain level is ≥ 4 on the visual analogue scale.
3. They have a sedentary lifestyle.

Exclusion Criteria:

1. Vaginismus requiring surgical treatment.
2. Any gynecological diseases such as pelvic organ prolapse, vulvar vestibulitis, vulvar pain, clitorodynia, vulvar dysesthesia, or any pelvic inflammatory diseases.
3. Lower urinary tract infection.
4. Husband with sexual dysfunction that prevents penetration.
5. Diseases involving nerves and muscles, such as myasthenia gravis.
6. Severe psychiatric disorder or cognitive relegation.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-20 (Estimated); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity. | Eight weeks
  The visual analogue scale (VAS): will be used to measure pain intensity for each woman in both groups. Each woman will be asked to mark the point on the scale that represents her pain level.
Quantification of pressure pain threshold in the perineum. | Eight weeks
  The pressure pain threshold in the perineum region will be evaluated with a pressure algometer.
Assessment of pelvic floor muscle tone. | Eight weeks
  It will be assessed by biofeedback perineometer.

SECONDARY OUTCOMES:
Measurement of cognition regarding vaginal penetration in women with lifelong vaginismus. | Eight weeks
  The Vaginal Penetration Cognition Scale (VPCQ) will be used to evaluate cognition regarding to vaginal penetration for all participants in both groups before and after the end of the treatment program.

CONTACTS AND LOCATIONS:
Overall Officials: Doaa A. Osman, PHD, Study Chair — Department of Women's Health, Faculty of Physical Therapy, Cairo University